CLINICAL TRIAL: NCT04740580
Title: Glutathione, Brain Metabolism and Inflammation in Alzheimer's Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Rajagopal V Sekhar, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: H48186
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Glycine; Acetylcysteine; Alanine

STUDY DESIGN:
Intervention Model Description: Placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glycine plus N-acetylcysteine (Experimental): Glycine and cysteine are amino-acid (protein) precursors of glutathione. Cysteine is provided as N-acetylcysteine
  Interventions: Dietary Supplement: Glycine; Dietary Supplement: N-acetylcysteine
- Alanine (Placebo Comparator): Alanine is an amino-acid (protein), and not a precursor of glutathione synthesis
  Interventions: Dietary Supplement: Alanine

INTERVENTIONS:
Dietary Supplement: Glycine — The active arm will supplement a combination of glycine and N-acetylcysteine (GlyNAC)
  Arms: Glycine plus N-acetylcysteine
Dietary Supplement: N-acetylcysteine — The active arm will supplement a combination of glycine and N-acetylcysteine (GlyNAC)
  Arms: Glycine plus N-acetylcysteine
Dietary Supplement: Alanine — The placebo arm will supplement Alanine
  Arms: Alanine

SUMMARY:
Alzheimer's disease (AD) is associated with significant, progressive cognitive decline. Key defects in mitochondrial fuel metabolism insulin resistance, inflammation and decreased brain glucose uptake are linked to AD. This trial will investigate the effects of supplementing glycine and N-acetylcysteine vs. alanine as placebo on these defects in AD, and examine the effects on cognition.

DETAILED DESCRIPTION:
Glutathione (GSH) deficiency, oxidative stress, mitochondrial dysfunction, insulin resistance and inflammation are linked to Alzheimer's disease (AD). In prior studies, investigators have shown that GSH deficiency contributes to mitochondrial impairment and oxidative stress, and that GSH deficiency can be corrected by supplementing its precursors glycine and cysteine (provided as N-acetylcysteine, NAC), with the combination termed GlyNAC.

This randomized clinical trial will evaluate the effect of GlyNAC vs. alanine placebo supplementation provided for 24-weeks to patients with AD, and measure changes in cognition, GSH concentrations, oxidative stress, brain glucose uptake, brain inflammation and insulin resistance.

Participants who are positive for a beta-amyloid PET scan and meeting cognitive screening criteria will be recruited, and enrolled only after meeting eligibility criteria. Before beginning study supplementation they will undergo imaging studies (MRI, FDG-PET and TSPO-PET scans), and only the FDG- and TSPO-PET scans will be repeated after completing 24-weeks of nutrient supplementation. Cognitive measurements, metabolic and mitochondrial measurements (as described below) will be done before supplementation, and after 12-weeks and 24-weeks of completing supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-85 years;
* Gradual and progressive memory loss for more than 1 year, with a Montreal Cognitive Assessment score of 10-20;
* Amyloid positivity on PET scan;
* Availability of a study partner.

Exclusion Criteria:

* hospitalization in past 3 months;
* use of insulin medications;
* untreated thyroid disease;
* creatinine levels >1.5 mg/dL;
* hemoglobin concentration <11.0 g/dL;
* known liver disease, or AST/ALT level >2x ULN;
* history of stroke, brain tumor, active heart failure or active cancer (removable basal cell cancers will not be an exclusion criteria);
* untreated depression or other severe psychiatric disorders;
* pregnancy or nursing (unlikely in this population)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognition | Day 0 of supplementation, and 12-weeks and 24-weeks after starting supplementation
  Measured using ADAS-Cog testing
Brain glucose uptake | Done before supplementation and 24-weeks after starting supplementation
  Measured using brain FDG-PET scan
Brain inflammation | Done before supplementation and 24-weeks after starting supplementation
  Done using brain TSPO-PET scan

SECONDARY OUTCOMES:
Activities of daily living | Day 0 of supplementation, 12-weeks and 24-weeks after starting supplementation
  Measured using the ADCS-ADL scale
Mitochondrial fuel oxidation | Day 0 of supplementation, 12-weeks and 24-weeks after starting supplementation
  Measured using indirect calorimetry in the fasted and post-glucose fed state
Red-blood cell glutathione, glycine, cysteine and glutamic aid | Day 0 of supplementation, 12-weeks and 24-weeks after starting supplementation
  Measured using UPLC
Oxidative stress | Day 0 of supplementation, 12-weeks and 24-weeks after starting supplementation
  Measured as plasma concentrations of TBARS and malondialdehyde
Damage due to oxidative stress | Day 0 of supplementation, 12-weeks and 24-weeks after starting supplementation
  Measured as plasma concentration of isoprostanes
Inflammatory cytokines | Day 0 of supplementation, 12-weeks and 24-weeks after starting supplementation
  Measured as plasma concentrations of IL6, TNFa
Endothelial dysfunction | Day 0 of supplementation, 12-weeks and 24-weeks after starting supplementation
  Measured as plasma concentrations of sICAM1, sVCAM1, E-selectin
Plasma concentration of Brain-derived neurotropic factor (BDNF) | Day 0 of supplementation, 12-weeks and 24-weeks after starting supplementation
  Measured using an ELISA kit
Mitochondrial energetics | Day 0 of supplementation, 12-weeks and 24-weeks after starting supplementation
  Measured using the Oroboros high-resolution respirometer

CONTACTS AND LOCATIONS:
Overall Officials: Rajagopal V Sekhar, M.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No